CLINICAL TRIAL: NCT06955559
Title: Magnesium Sulfate in Bronchial Asthma and Acute Bronchiolitis in Children
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Ibrahim Mostafa, residant doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mg bronchialasthma bronchiolis
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- study group (Active Comparator): All children more than 1 month and less than 18 year cases with bronchial asthma and acute bronchiolitis.
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate — inhaled magnesium sulfate (MgSO4)

SUMMARY:
Asthma is a prevalent disease that affects as many as334 million individuals worldwide, and is a major source of disability and premature death in children(1).

Asthma affects 7.1 million children in the United States (2). and is the most common pediatric chronic disease(3).Globally, the prevalence of pediatric asthma varies from 10% to 30%. Its symptoms range from chronic cough to life-threatening bronchospasm.(4,5,6).The most common triggers of asthma exacerbations in both younger and older children are viral respiratory tract infections, exposure to allergens, tobacco smoke, air pollutants, cold or dry air, and poorly controlled asthma(4,7).Current management strategies for acute asthma recommend a stepwise approach, with first-line standard therapy followed by additional therapeutic options(8).Firstline therapy consists of inhaled rapid-acting selective b2-agonists, inhaled ipratropium bromide, and oral or intravenous corticosteroids. Response to standard acute asthma therapy is variable, influenced by factors that cannot be assessed or accounted for urgently such as genetic polymorphisms(9-12).For patients who do not respond adequately to first-line therapy, further improvement can be seen with additional therapy such as inhaled magnesium sulfate (MgSO4) or intravenous aminophylline, terbutaline, or magnesium sulfate. Though all available second-line therapeutic agents produce bronchodilatory effects, magnesium sulfate produces fewer side effects, is more widely available, and costs less than other second-line therapies(13). This combination of efficacy, few side effects, wide availability, and low cost suggest that magnesium sulphate is a promising therapeutic agent that deserves further consideration for use in children with acute asthma. Acute bronchiolitis (AB) is an infection of the lower respiratory tract that is caused by viral agents, especially respiratory syncytial virus, most prevalent in children aged less than 24months(14). It is the most common reason for hospital admissions in the first year of life, representing a significant health burden worldwide. Bronchiolitis usually demonstrates a benign course, most patients are treated as outpatients but progression to severe illness may occur rapidly and respiratory support and admission to pediatric intensive care unit (PICU) may be required promptly in some cases(14). It is characterized by damage of epithelial cells leading to ciliary destruction, airway inflammation, edema, and increased mucus production. Mucus plugs and cellular debris obstruct bronchiolar lumens and result in various degrees of respiratory distress(15). Current recommendations for treatment of AB focus on supportive care, including respiratory support, oxygen supplementation if needed, and adequate hydration. Other treatment agents, such as bronchodilators, hypertonic saline, corticosteroids, and antiviral/antibacterial agents, showed no clearly defined benefit. Only highflow nasal cannula (HFNC) oxygen therapy has been elucidated as a new and promising tool for respiratory support for these patients(16-23).

* Magnesium sulfate was also investigated as a treatment option for bronchiolitis in few studies

ELIGIBILITY:
Inclusion Criteria:

* All children more than 1 month and less than 18 years cases with bronchial asthma and acute bronchiolitis

Exclusion Criteria:

* All children less than 1 month and more than 18 years congenital heart disease

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Safty of intravenous magnesium sulfate | baseline
  Safty of intravenous magnesium sulfate is defined as development of serious adverse events such as hypotension requiring medical intervention.